CLINICAL TRIAL: NCT04327778
Title: Automate Music Therapy for the Management of Behavioral Disorders in Nursing Homes
Acronym: MAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-AOI-09
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Alzheimer Disease; Major Neurocognitive Disorder
MeSH Terms: conditions — Alzheimer Disease | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music therapy (Experimental): Patients will be exposed every two weeks
  Interventions: Procedure: Music Therapy

INTERVENTIONS:
Procedure: Music Therapy — Automate music therapy every two weeks

SUMMARY:
Alzheimer disease is the most common neurodegenerative brain disease that causes cognitive impairment in the elderly but also behavioral and psychological symptoms. Among these symptoms, agitation is one of the most dangerous because it put the patient and their caregivers in danger. Sleep disorders can be the cause of many psychiatric symptoms leading directly or indirectly to agitation. Music therapy is the non-drug therapy which has been shown to be the most effective in managing agitation and sleep disorders. With the MAGE protocol, the investigators propose to take care of behavioral disorders in severe Alzheimer patients living in nursing home through sequences of music therapy (stimulation, relaxation) automatically initiated by an actigraph that will detect sleep disorders. These subjects will be exposed for 2 weeks over a month. Behavioral and sleep disorders will be evaluated objectively by actigraphy but also by standardized scales, as the others neuropsychiatric symptoms found classically in this disease. Thanks to this project, the investigators hope to improve the quality of life of these patients by preventing them from putting themselves in danger, by reducing their neuropsychiatric symptoms and their use of medication, which has often deleterious side effect and also by reducing the workload of caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years old
* Male or Female
* Patients with a diagnosis of Alzheimer disease according to the criteria of NINCDS-ADRDA or typical or atypical Alzheimer disease
* MMSE < 20
* Patient residing in nursing home
* Voluntary, written and informed consent of the patient himself or its legal representative (guardian/curator)
* Affiliation to a social security system

Exclusion Criteria:

* Prescription of a new psychotropic treatment (hypnotic, anxiolytic, antidepressant, antipsychotic) in week prior to the evaluation
* Hearing loss preventing the patient from responding perfectly to the therapeutic solutions provided

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric tests scores | At 3 months
  NeuroPsychiatric Inventory before exposure and at the end of each exposure, score from 0 to 120
Nightly agitation | At 3 month
  The number of movements of the patient by the actigraphy, before exposure and at the end of each exposure

SECONDARY OUTCOMES:
Number of falls | At 3 months
  Number of falls by actigraphy
Sleeping troubles | At 3 months
  Hours of sleep by actigraphy
Rate of anxiety | At 3 months
  Anxiety rate measured by taking anxiolytic drugs

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France